CLINICAL TRIAL: NCT05865444
Title: Prevention of Eating Habits Associated With Obesity in Adolescents Through a Wise Intervention
Brief Title: Prevention of Eating Habits Associated With Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Deusto (Other)
Responsible Party: Principal Investigator, Esther Calvete, Principal Investigator, Deusto Stress Research Team, University of Deusto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ETK-43/21-22
Record Dates: First submitted 2023-02-20; First posted 2023-05-18 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Obesity, Adolescent; Eating, Healthy
Keywords: Adolescence; Prevention; Healthy food intake; Unhealthy food intake; Wise intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with two groups will be used. Randomization will be done by clusters, using the classroom as the unit. First, the schools will be selected according to their characteristics. Then, for each school and grade, half of the classrooms will be randomly assigned to the experimental condition (values alignment condition) and the other half to the active control condition (traditional educational intervention) in parallel for the duration of the study.
Who Masked: Participant, Outcomes Assessor
Masking Description: Allocation will be concealed to the participants and teachers. Assessment will be done online through self-reports.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Values alignment wise intervention (Experimental): 1 hour wise intervention (based on a values alignment approach) consisting on several tasks (online and paper-based tasks) to be completed individually.
  Interventions: Behavioral: Values alignment wise intervention
- Traditional educational intervention (Active Comparator): 1 hour traditional educational intervention on nutrition and physical exercise. This will also include reading and writing exercises.
  Interventions: Behavioral: Educational traditional intervention

INTERVENTIONS:
Behavioral: Values alignment wise intervention — The intervention includes: (1) reading materials, such as recent journalistic works that expose the deceptive and manipulative marketing practices of food companies and the harmful effects of these practices on society, with particular emphasis on harm to young children and the economically disadvantaged. Stories from other young people will also be included in order to contribute to the perception of widespread outrage and to suggest how that outrage can be channeled into taking a stand against the injustice perpetrated by food companies by eating less unhealthy or healthier food; (2) writing exercises, such as a story with a brief statement of what the participants would tell a younger child about the ads; and (3) an interactive activity, called "Make It Real" in which they are shown pictures of food ads and allowed to write and draw about them, making whatever changes (e.g., crossing out and substituting words) they feel necessary to make the ad "real" (i.e., no longer misleading).
  Arms: Values alignment wise intervention
Behavioral: Educational traditional intervention — The educational intervention includes information on nutrition and physical exercise. It includes reading and writing exercises.
  Arms: Traditional educational intervention

SUMMARY:
This study evaluates the effectiveness of a Wise Intervention based on a values alignment approach to improve obesity-related eating habits in Spanish adolescents. Half of the participants will receive the experimental intervention, while the other half will receive a control intervention.

DETAILED DESCRIPTION:
Obesity in adolescence is associated with physical and mental health problems and predicts obesity in adulthood. Adolescence may be an ideal time to target interventions, as this is when numerous health-related habits are consolidated. Several universal preventive interventions have been carried out in educational centers for the promotion of healthy eating habits. However, the results of reviews and meta-analyses have concluded that most are not cost-effective for producing long-term changes in the dietary preferences of young people. The so-called wise interventions paradigm is an innovative approach to interventions that involve a set of rigorous techniques grounded in research to help people improve in a variety of life settings. Recently, it has been developed a wise intervention aimed at improving adolescents' daily dietary choices. This intervention, called the values alignment intervention, focused on the role of marketing on the behavior of children and adolescents who are exposed to a relentless barrage of marketing from the food industry. The values alignment intervention seeks to neutralize the positive emotional associations with junk food that marketing generates and presents the rejection of unhealthy foods in favor of healthy alternatives as a way to live up to two values that are important to adolescents: (1) the desire to be autonomous from adult control, and (2) the desire for social justice. In two randomized controlled trials, it has been demonstrated that the intervention reduced implicit positive associations with junk food and substantially improved dietary choices, especially in boys. In addition, there were significant differences in attitudinal variables related to healthy eating. These promising results suggest that reframing unhealthy eating as incompatible with important youth values could be a low-cost solution to produce changes in adolescent attitudes and dietary choices. Therefore, the general objective of this project is to adapt the values alignment intervention to improve obesity-related eating habits in Spanish adolescents and evaluates its effectiveness. It is therefore a highly innovative project with great potential for social impact in the field of health promotion.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by the adolescents and their parents.
* To be fluent in Spanish and/or Euskera.

Exclusion Criteria:

* Lack of permission by parents and the adolescent.
* Lack of understanding of the instructions.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 591 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline scores of healthy and unhealthy food intake using the questionnaire developed by Stok et al. (2015). | Baseline, 1 week, 3 months
  It consists of four items that ask frequency of consumption of healthy and unhealthy food. It provides an index of unhealthy eating. Five response categories are provided: "none", "1", "2", "3", "4", or "more than 4 per day".
Change from baseline scores of body mass index. | Baseline, 3 months
  Self-reported height (cm) and weight (kg) for BMI calculation.

SECONDARY OUTCOMES:
Change from baseline scores of the alignment of healthy eating habits with the values of adolescents using a questionnaire developed from Bryan et al. (2019). | Baseline, 1 week, 3 months
  It consists of seven items that assess adolescents' interpretation of healthy eating as addressing social justice issues (4 items) and as an assertive behavior expressing autonomy and independence (3 items). Each item is scored 0-4 (0 = not true; 4 = extremely true), yielding a total between 0 and 28.
Change from baseline scores of the social attractiveness of healthy eating using a questionnaire developed by Bryan et al. (2019). | Baseline, 1 week, 3 months
  It consists of three items that assess social attractiveness of healthy eating. Each item is scored 0-4 (0 = not at all agree; 4 = totally agree), yielding a total between 0 and 12.

CONTACTS AND LOCATIONS:
Overall Officials: Esther Calvete, PhD, Principal Investigator — University of Deusto
Locations (1):
- University of Deusto, Bilbao, Vizcaya, Spain

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be available at OSF when the results of the study are published.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The study protocol and informed consent protocol will be published at clinicaltrials.org Data will be available at OSF when the results are published.
Access Criteria: Public

REFERENCES:
- [Background] Ashton LM, Sharkey T, Whatnall MC, Williams RL, Bezzina A, Aguiar EJ, Collins CE, Hutchesson MJ. Effectiveness of Interventions and Behaviour Change Techniques for Improving Dietary Intake in Young Adults: A Systematic Review and Meta-Analysis of RCTs. Nutrients. 2019 Apr 11;11(4):825. doi: 10.3390/nu11040825. PMID 30979065
- [Background] Bryan CJ, Yeager DS, Hinojosa CP. A values-alignment intervention protects adolescents from the effects of food marketing. Nat Hum Behav. 2019 Jun;3(6):596-603. doi: 10.1038/s41562-019-0586-6. Epub 2019 Apr 15. PMID 30988478
- [Background] Bryan CJ, Yeager DS, Hinojosa CP, Chabot A, Bergen H, Kawamura M, Steubing F. Harnessing adolescent values to motivate healthier eating. Proc Natl Acad Sci U S A. 2016 Sep 27;113(39):10830-5. doi: 10.1073/pnas.1604586113. Epub 2016 Sep 12. PMID 27621440
- [Background] Kobes A, Kretschmer T, Timmerman G, Schreuder P. Interventions aimed at preventing and reducing overweight/obesity among children and adolescents: a meta-synthesis. Obes Rev. 2018 Aug;19(8):1065-1079. doi: 10.1111/obr.12688. Epub 2018 Apr 19. PMID 29671938
- [Background] Stok FM, de Vet E, de Wit JB, Luszczynska A, Safron M, de Ridder DT. The proof is in the eating: subjective peer norms are associated with adolescents' eating behaviour. Public Health Nutr. 2015 Apr;18(6):1044-51. doi: 10.1017/S1368980014001268. Epub 2014 Jun 18. PMID 24940622
- [Background] Walton GM, Wilson TD. Wise interventions: Psychological remedies for social and personal problems. Psychol Rev. 2018 Oct;125(5):617-655. doi: 10.1037/rev0000115. PMID 30299141

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT05865444/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT05865444/ICF_001.pdf